CLINICAL TRIAL: NCT01653119
Title: Peking and Rotterdam on Mission to Reduce Coronary Artery Disease
Acronym: PROMISS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Wei Gao, doctor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUCRP-004
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-03

CONDITIONS: Acute Coronary Syndrome; Diabetes Mellitus
Keywords: Acute coronary syndrome; Diabetes mellitus; Statins; High loading dose; Recurrent events
MeSH Terms: conditions — Acute Coronary Syndrome; Diabetes Mellitus | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High loading dose of rosuvastatin (Active Comparator): rosuvastatin 20mg/d×1w
  Interventions: Drug: Rosuvastatin
- Routine rosuvastatin therapy (Active Comparator): rosuvastatin 10mg/d×1w
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Both of the two groups will be given standard ACS treatment according to treatment guidelines during the following 1 year.
  Other Names: Crestor

SUMMARY:
The purpose of this study is to explore the effect of 20mg high loading dose of rosuvastatin on recurrent events in patients with established DM who is admitted for an ACS.

ELIGIBILITY:
Inclusion Criteria:

* • Men or women ≥40 years of age admitted with a clinical diagnosis of ACS. The diagnosis should be based on the combination of typical ischemic chest complaints and objective evidence of myocardial ischemia or myocardial necrosis as demonstrated by the electrocardiogram (ECG) or elevated cardiac markers, as follows:
* Typical ischemic chest pain, lasting 10 minutes or more, within the preceding 24 hours, AND either
* ECG changes indicative of myocardial ischemia within 24 hours after the onset of chest pain (ECG showing persistent or non-persistent ST-segment elevation >1.0 mm in two or more contiguous leads or dynamic ST-segment depression >1.0 mm in two or more contiguous leads) or
* Elevated biomarkers of myocardial necrosis within 24 hours after the onset of chest pain (i.e. CK-MB >1 times the upper limit of normal of the local laboratory, or Troponin-T >0.1 ng/ml.

  * A diagnosis of DM type II prior to the index ACS
  * Written informed consent

Exclusion Criteria:

* • Myocardial ischemia precipitated by a condition other than atherosclerotic coronary artery disease (e.g. arrhythmia, severe anemia, hypoxia, thyrotoxicosis, cocaine, severe valvular disease, hypotension).

  * Severely-impaired left ventricular function (ejection fraction <30%) or end-stage congestive heart failure NYHA-class III or IV (in order to avoid lost-to-follow-up due to non-acute coronary syndrome events).
  * Severe chronic kidney disease with measured or calculated glomerular filtration rate (Cockgroft-Gault or MDRD4 (Modification of Diet in Renal Disease) formula) of <30 ml/min/1.73m2, or renal dialysis.
  * Co-existent condition associated with a life-expectancy <12 months, or otherwise unlikely to appear at all scheduled follow-up visits.
  * Known serious or hypersensitivity reactions to HMG-CoA reductase inhibitors.
  * Triglyceride (TG) level ≥500 mg/dL (5.65 mmol/L) at screening, because patients with very high triglyceride levels warrant treatment with agents that may increase the risk of side effects associated with statin drugs.
  * Active liver disease or hepatic dysfunction, as determined by alanine aminotransferase (ALT [SGPT]) >3 x ULN or bilirubin levels >1.5 x ULN at screening.
  * Myopathy.
  * Not using effective contraceptive methods.
  * Participation in any investigational drug study less than 30 days prior to enrolment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2012-04; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
A composite of cardiovascular mortality or a clinical diagnosis of a non-fatal ACS | during 12 months follow-up

SECONDARY OUTCOMES:
A composite of cardiovascular mortality or a clinical diagnosis of a non-fatal ACS | during 30 days follow-up

OTHER OUTCOMES:
The proportion of any AST or ALT >3 x ULN or CK >5 x ULN | during the 1-year follow up period

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China